CLINICAL TRIAL: NCT04681599
Title: Comparison of Different Modalities in Reducing Airborne Particulate Concentrations During Aerosol Generating Procedures for Health Volunteers: a Randomized Cross-over Trial
Brief Title: Different Modalities in Reducing Airborne Particulate Concentrations During AGP for Health Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: AGP aerosol 002
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Transmission, Patient-Professional
Keywords: aerosol generating procedure; high-flow nasal cannula; nebulization; aerosol therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Nebulization without filter or scavenger (No Intervention): Subject will use a standard nebulizer
- Nebulization with a filter or scavenger (Experimental): Subject will use a nebulizer with a filter placed at the other end of nebulizer mouthpice or a scavenger outside the nebulizer mask
  Interventions: Device: Filter; Device: Scavenger face tent
- High-flow nasal cannula (No Intervention): Subject will use high-flow nasal cannula at 40 L/min
- High-flow nasal cannula with a scavenger face tent (Experimental): Subject will use high-flow nasal cannula at 40 L/min, with a scavenger face tent
  Interventions: Device: Scavenger face tent
- High-flow nasal cannula with a surgical mask (Active Comparator): Subject will use high-flow nasal cannula at 40 L/min, with a surgical mask over nasal cannula
  Interventions: Device: Filter

INTERVENTIONS:
Device: Filter — Filter is used to capture any individual bacteria or viruses that might be suspended within inhaled or exhaled gases
  Arms: High-flow nasal cannula with a surgical mask; Nebulization with a filter or scavenger
Device: Scavenger face tent — A face tent is connected to a vacuum resource to continuously suction the exhaled gas from the subject, in order to reduce the transmission risk of virus or bacteria
  Arms: High-flow nasal cannula with a scavenger face tent; Nebulization with a filter or scavenger

SUMMARY:
Several clinical procedures have been described as aerosol generating procedure (AGP), including nebulization, high-flow nasal cannula oxygen therapy, noninvasive ventilation, and bronchial hygiene treatment, etc. However, the understanding on the transmission risk of these treatments is still unclear, particularly the methods to reduce the airborne particulate concentrations during these treatments are still lacking. This study is aimed to compare different modalities in reducing airborne particulate concentrations during these aerosol generating procedures, in order to find the most effective method to reduce particle concentrations, ultimately to decrease the transmission risk and protect health care providers.

ELIGIBILITY:
Inclusion Criteria:

• Ages 18-65, Male or Female

Exclusion Criteria:

* Chronic lung disease, including asthma, COPD, etc.
* Upper airway anatomical abnormities
* Pregnancy
* Uncontrolled Diabetes, hypertension, or untreated thyroid disease
* Has any of the following symptoms in the last 21 days: sore throat, cough, chills, body aches for unknown reasons, shortness of breath for unknown reasons, loss of smell, loss of taste, fever at or greater than 100 degrees Fahrenheit.
* COVID-19 test positive within 21 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
aerosol particle concentrations at 1 foot away from subject's face | 5 mins
  aerosol particle concentrations will be recorded continuously for 5 mins during the use of each device at 1 foot away from subject's face
aerosol particle concentrations at 3 feet away from subject's face | 5 mins
  aerosol particle concentrations will be recorded continuously for 5 mins during the use of each device at 3 feet away from subject's face

SECONDARY OUTCOMES:
subject's comfort | 5 minutes after using the device
  subject's comfort will be self-evaluated using a visual numerical scale (VNS) ranging between 1 (very uncomfortable) and 5 (very comfortable)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, PhD, Principal Investigator — Rush University
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
individual participant data would not be shared

REFERENCES:
- [Result] Dhand R, Li J. Coughs and Sneezes: Their Role in Transmission of Respiratory Viral Infections, Including SARS-CoV-2. Am J Respir Crit Care Med. 2020 Sep 1;202(5):651-659. doi: 10.1164/rccm.202004-1263PP. No abstract available. PMID 32543913
- [Result] Li J, Fink JB, Ehrmann S. High-flow nasal cannula for COVID-19 patients: low risk of bio-aerosol dispersion. Eur Respir J. 2020 May 14;55(5):2000892. doi: 10.1183/13993003.00892-2020. Print 2020 May. PMID 32299867
- [Result] Fink JB, Ehrmann S, Li J, Dailey P, McKiernan P, Darquenne C, Martin AR, Rothen-Rutishauser B, Kuehl PJ, Haussermann S, MacLoughlin R, Smaldone GC, Muellinger B, Corcoran TE, Dhand R. Reducing Aerosol-Related Risk of Transmission in the Era of COVID-19: An Interim Guidance Endorsed by the International Society of Aerosols in Medicine. J Aerosol Med Pulm Drug Deliv. 2020 Dec;33(6):300-304. doi: 10.1089/jamp.2020.1615. Epub 2020 Aug 12. PMID 32783675
- [Result] Kaur R, Weiss TT, Perez A, Fink JB, Chen R, Luo F, Liang Z, Mirza S, Li J. Practical strategies to reduce nosocomial transmission to healthcare professionals providing respiratory care to patients with COVID-19. Crit Care. 2020 Sep 23;24(1):571. doi: 10.1186/s13054-020-03231-8. PMID 32967700